CLINICAL TRIAL: NCT06519812
Title: Efficacy and Safety of Endoscopic Combined Intrarenal Surgery vs. Percutaneous Nephrolithotomy for Treatment of Staghorn Calculi, A Prospective Randomized Study
Brief Title: Endoscopic Combined Intrarenal Surgery vs. Percutaneous Nephrolithotomy for Treatment of Staghorn Calculi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Maher Mohamed Abdelrehem Mohamed, Assistant Lecturer of Urology Faculty of Medicine, Al-Azhar University (Damietta), Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Urosurg./MD/2023/0008
Record Dates: First submitted 2024-06-27; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Urinary Calculi
MeSH Terms: conditions — Urinary Calculi | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Group I (PCNL group) (Experimental): 50 patients will undergo percutaneous nephrolithotomy (PCNL).
  Interventions: Procedure: Combined Intrarenal Surgery and percutaneous nephrolithotomy
- Group II (ECIRS group) (Experimental): 50 patients will undergo endoscopic combined intrarenal surgery (ECIRS).
  Interventions: Procedure: Combined Intrarenal Surgery and percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Combined Intrarenal Surgery and percutaneous nephrolithotomy — A study was conducted to compare endoscopic combined intrarenal surgery and percutaneous nephrolithotomy as modalities of treatment for staghorn stones.

SUMMARY:
This is a prospective randomized study to compare endoscopic combined intrarenal surgery and PCNL as modalities of treatment for staghorn stones. In terms of efficacy and safety

DETAILED DESCRIPTION:
This is a prospective randomized study to compare endoscopic combined intrarenal surgery and PCNL as modalities of treatment for staghorn stones. In terms of efficacy and safety The efficacy will be studied at stone-free rate While efficacy will be studied using DMSA scan pre- and post-procedures in addition to the safety of each procedure with regard to intra- and post-operative complications,.

ELIGIBILITY:
Inclusion Criteria:

* Patients are more than 18 and less than 65 years old.
* Patients with renal staghorn stones based on imaging modalities (stones occupying the renal pelvis and extending into at least 2 major calyces).

Exclusion Criteria:

* Patients with renal insufficiency (serum creatinine > 1.6 mg/dl)
* patients with active urinary tract infection.
* Patients with congenital renal anomalies.
* Morbid obesity (BMI > 35 kg/m2).
* Pregnancy.
* Bleeding Coagulopathy.
* Skeletal deformity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
stone-free rate | 3 months postoperative
  Stone-free is defined as no residual stones on CT-UT or clinically insignificant residual fragments (CIRF) less than 4 mm in diameter.
  It will be measured twice, first immediately postoperatively, and then again after 3 months of the procedure.

SECONDARY OUTCOMES:
Safety of the procedure | intraoperative, early (in the first day postoperative) and late complications (3 months after the surgery).
  Intra and post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Maher Abdelrehem Mohamed, Master, Principal Investigator — assistant lecturer of urology , Al-Azhar University (Damietta)
Locations (1):
- Al-Azhar University Hospital (New Damietta), Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No